CLINICAL TRIAL: NCT02507063
Title: Determining the Correlation of Optic Nerve Sheath Diameter With Intracranial Pressure in Children
Brief Title: Optic Nerve Sheath Diameter and Intracranial Pressure (ICP) in Children
Status: Withdrawn | Type: Observational
Sponsor: Anna Rominger (Other)
Responsible Party: Sponsor-Investigator, Anna Rominger, Assistant Professor, University of Louisville
Organization: University of Louisville (Other)
Other Study IDs: 15.0326
Record Dates: First submitted 2015-07-18; First posted 2015-07-23 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Intracranial Hypertension
MeSH Terms: conditions — Intracranial Hypertension | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- study subjects: Patients age 0-18 with intracranial monitoring devices in place or requiring a VP shunt revision who receive a ocular ultrasound evaluating ONSD
  Interventions: Procedure: ultrasound

INTERVENTIONS:
Procedure: ultrasound — Ocular ultrasound to look at the optic nerve sheath diameter in patients with an intracranial monitoring device or with a ventriculoperitoneal shunt malfunction requiring revision

SUMMARY:
The use of optic nerve sheath diameter (ONSD) measurements as a non invasive test for raised ICP has many potential benefits. This includes having assessments that can be made at the bedside instead of requiring patient transport to CT or MRI, which in itself can cause a rise in ICP. If ONSD represents an acute and sensitive measurement of elevated ICP, it may prove useful in the emergency department (ED) setting in the evaluation of shunts used for cerebrospinal fluid (CSF) diversion. The investigators hypothesize that ONSD will correlate with measured ICP and thus be a reliable tool for the bedside assessment of ICP. The investigators further hypothesize that ONSD changes will correlate with changes in ICP, making it a useful bedside tool for assessing ICP changes over time. This is a prospective, observational study using a convenience sample. Children who are 0 - 18 years old who have an invasive intracranial ICP monitoring device admitted to the hospital Pediatric Intensive Care Unit (PICU) are eligible for participation in the study. Children who are 0-18 years old who are determined to require a shunt revision following evaluation in the ED will also be included in the study. 10. After the invasive intracranial pressure monitoring device is placed, for every recruited patient, ONSD measurements will be taken and the ICP will be recorded 8 hours post placement and then repeated 3 times a day until the intracranial pressure monitoring device is removed.12. For ventriculoperitoneal (VP) shunt revision patients, the investigators will obtain a measurement just before surgery, immediately post-op, and then 12 hours, 24 hours, and 36 hours post-op. If the patient is otherwise ready for discharge prior to 36 hours, the measurement may be omitted or done early so as to not unnecessarily prolong the hospitalization

ELIGIBILITY:
Inclusion Criteria:

* Children between 0 years and 18 years of age
* Children who are determined to need an invasive intracranial monitoring device in the ED and admitted to the PICU
* Children who undergo VP shunt revisions at the study site

Exclusion Criteria:

* Children with an invasive intracranial monitoring device that is malfunctioning
* Prior adverse reactions to ultrasound gel
* Pre-existing ophthalmologic conditions that could cause a baseline increase in ONSD, including glaucoma or severe ocular trauma
* Children with ocular or facial trauma that would impede ONSD measurements

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who are 0 - 18 years old who have an invasive intracranial ICP monitoring device admitted to PICU and children who are 0-18 years old who are determined to require a shunt revision following evaluation in the ED.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
The correlation (composite of multiple measurements) of ONSD measurements by sonography in patients with intracranial pressure measurements by invasive intracranial monitors. | 3 years

SECONDARY OUTCOMES:
ONSD measurements by sonography in patients with VP shunt malfunction as evidenced by CT scan | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anna H Rominger, MD MPH MsC, Study Director — University of Louisville

IPD SHARING:
Plan to Share IPD: No